CLINICAL TRIAL: NCT06486220
Title: PFLL Combined With PD-1 Antibody With or Without FMT for Oligometastatic NPC,a Phase III ,Open, Randomized Clinical Trial.
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yun-fei Xia (Other)
Responsible Party: Sponsor-Investigator, Yun-fei Xia, Sun Yat-sen University Cancer Prevention Center, Sun Yet-Sen University Cancer Center
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-FXY-120
Record Dates: First submitted 2024-06-21; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flora Transplantation group (Experimental): 5-Fu+DDP+anti-PD-1 mAb+FMT
  Interventions: Drug: Intestinal bacteria freeze-dried powder capsules
- Control group (No Intervention): 5-Fu+DDP+anti-PD-1 mAb

INTERVENTIONS:
Drug: Intestinal bacteria freeze-dried powder capsules — Oral healthy intestinal bacteria freeze-dried powder capsules, tid
  Other Names: 5-FU+DDP+anti-PD-1 mAb
  Arms: Flora Transplantation group

SUMMARY:
There is a correlation between gut microbiota and immunotherapy reactivity, and regulating gut microbiota through FMT can prevent primary resistance to immune checkpoint inhibitors and further improve the effectiveness of tumor immunotherapy.Therefore, on the basis of previous studies, this study intends to explore whether intestinal flora transplantation can improve the anti-tumor efficacy of low-dose long term 5-FU pumping ("old fire soup") therapy combined with immunotherapy and reduce the occurrence of toxic side effects in patients with metastatic nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
Experimental group (PFLL + PD-1 + FMT) :

5-Fu 200mg/ m2 /d, D1-30 + cisplatin 80mg/ m2, d1, 28 or D1-3, 28-30 + triplizumab 240mg, d1, 22 + FMT 10 capsules in the morning, middle and evening, D-5-3, 11-13, 38-40;Every 60 days/cycle, PFLL + PD-1 + FMT is given for a maximum of 6 cycles.

Control group (PFLL + PD-1) :

5-Fu 200mg/ m2 /d, D1-30 + cisplatin 80mg/ m2, d1, 28 or D1-3, 28-30 + triplizumab 240mg, d1, 22;PFLL + PD-1 is given a maximum of 6 cycles per 60 days/cycle.

ELIGIBILITY:
Inclusion Criteria:

1. 18-60 years old;
2. Pathological diagnosis of nasopharyngeal carcinoma;
3. Patients diagnosed with oligometastatic nasopharyngeal carcinoma who meet stage IVb as defined by the International Union against Cancer and the American Joint Committee on Cancer (UICC/AJCC) staging System (8th edition) (Oligometastatic as ≤3 organs and ≤5 sites of metastasis);
4. Patients with metastatic nasopharyngeal carcinoma who had not previously received systematic chemotherapy for the disease in this study, except neoadjuvant chemotherapy, concurrent chemoradiotherapy or adjuvant chemotherapy received 6 months before the first administration;
5. Karnofsky's functional status score should be at least 70 points (if the functional status score is decreased due to tumor, it should be appropriately relaxed after the researchers' judgment, and the minimum score should be no less than 50 points, as shown in Annex I);
6. According to the RECIST1.1 evaluation criteria, there should be at least 1 measurable lesion, and the measurable lesion should not have received local treatment such as radiotherapy;
7. Expected survival ≥3 months;
8. A tolenrant organs.

Exclusion Criteria:

1. allergy to 5-FU, gemcitabine, cisplatin, other monoclonal antibodies, or any component of triplimab
2. Prior treatment with PD-1 receptor or its ligand PD-L1 or cytotoxic T lymphocyte-associated protein 4 (CTLA4) receptor;
3. Had major surgery other than diagnosis of nasopharyngeal cancer within 28 days prior to randomization or was expected to require major surgery during the study period;
4. Patients with severe damage of intestinal barrier such as sepsis, active massive bleeding of digestive tract and perforation due to various reasons;
5. Currently diagnosed with fulminant colitis or toxic megacolon;
6. Enteral nutrition patients who cannot tolerate 50% of heat calorie requirements due to severe diarrhea, significant fibrous intestinal stenosis, severe gastrointestinal bleeding, high-flow intestinal fistula, etc.;
7. patients with any active autoimmune disease or a history of autoimmune diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 1-year PFS 40%
  Progression-free survival

SECONDARY OUTCOMES:
OS | 24 months
  overall survival

IPD SHARING:
Plan to Share IPD: No